CLINICAL TRIAL: NCT03367650
Title: Epidemiology and Genetics of the Amyotrophic Lateral Sclerosis in the French West Indies
Acronym: SLA-DOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBM-PAP-2013/55
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; epidemiology; genetic; environmental factor
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Bi-centric epidemiological prospective, cross-sectional descriptive study coupled with a longitudinal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALS's patients in Guadeloupe and Martinique (Other): We shall determine:
  * Impact of ALS in Guadeloupe and Martinique
  * Prevalence of the ALS in Guadeloupe and Martinique on the duration of the study
  * The distribution of ALS various phenotypes in our population of patients.
  * We shall collect the date of the beginning of the symptoms of the SLA, the date of diagnosis of ALS, the date of death for the same individual and the origin of the death, the weight, the size, the albumin, CRP; in order to establish the forecast of the various clinical forms, the description of the evolution of the nutritional state.
  * Search for transfers of genes TARDBP, VCP, SOD1 known and involved in the disease
  * Search for possible environmental factors
  Interventions: Dietary Supplement: Blood sample and environmental survey

INTERVENTIONS:
Dietary Supplement: Blood sample and environmental survey — The intervention corresponds to a 10 ml of Blood sample and an environmental survey.

SUMMARY:
The diagnosis and the follow-up of the patients reached of SLA is centralized, since a few years, at the the Caribbean Reference center of the rare neurological diseases (CERCA labélisé in 2006) in Martinique and at the Unity of coverage of the neuromuscular Diseases, SLA and the rare neurological diseases (create in 2010) in Guadeloupe. Several phenotypic characteristics seemed to us to take out again data collected during the follow-up of the patients (26 in Guadeloupe, since the creation of the unity) in particular patients' high proportion of exceptionally long evolution (more than 10 years). Besides, we diagnosed several cases (10 cases in Guadeloupe since 2000) of association SLA- Parkinsonien Syndrome.

This association, considered as exceptional could establish a particular phenotypic entity which we would like to describe. We are interested also originally geographical of the patients, with the hypothesis that he could exist in the Antilles one or several geographical isolates of the disease allowing to lead a étiologique investigation in search of a possible genetic or environmental cause.

DETAILED DESCRIPTION:
The amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterized by progressive muscular paralysis due to degeneration of motor neurons in the primary motor cortex, corticospinal pathway, brain stem and spinal cord. The incidence is estimated at 2/100 000 per year and prevalence at approximately 4/100000.

Various clinical forms are described. The disease is fatal is 3-5 years on average.

The majority of cases are sporadic and of unknown origin but 5-10% are familial and present for 20% of them, mutations in the SOD1 (21q22.11) gene. Other genes have recently been implicated in ALS. Environmental toxic factors have been extensively researched. Beta-methylamino-L-alanine (BMAA), a neurotoxic nonprotein amino acid produced by most cyanobacteria, has been proposed to be the causative agent of the ALS-Parkinsonism Complex on the island of Guam in the Pacific Ocean.

Epidemiology and clinical features of ALS have never been studied in Caribbean countries.

The main purpose of the study will be to evaluate the incidence of ALS in Guadeloupe and Martinique.

Secondary purposes will be:

1. to evaluate the presence of specific phenotypic features;
2. to establish he prognosis of different clinical forms;
3. to study the genes implicated in ALS and quantify theexposure to BMAA.

Since 2000, the diagnosis of ALS is made in about 20 patients per year in Guadeloupe and Martinique(for a total population of 800000 inhabitants) but the incidence and the clinical presentation of ALS in the French West Indiesare unknown.

The exceptional association of ALS and parkinsonism is regularly observed in Guadeloupe. We propose to perform a prospective descriptive and longitudinal epidemiological study to determine the incidence of ALSin the French West Indies. In parallel we will study the involvement of genetic andenvironmental toxic factors as etiological factor for this disease.

Primary outcome:

- the impact of ALS in Guadeloupe and Martinique

Secondary outcomes:

* Assess the clinical characteristics (presence of phenotypic features?),
* the prognosis of different clinical forms study,
* to establish the genetic factors of the ALS and to search potential environmental factors

ELIGIBILITY:
Inclusion Criteria:

* Patient or third-party responsible for receiving information on the study and who signed informed consent ;
* Patient age over 18 years;
* Patient living in the Antilles;
* Patient with ALS or SLP (primary lateral sclerosis, pure central form of ALS).

Exclusion Criteria:

* Patient non-affiliated to the social security scheme ;
* in case of difficulty of monitoring patient, exclusion of the longitudinal study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-05-13 (Actual); Primary Completion 2020-05-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
the impact of amyotrophic lateral sclerosis in Guadeloupe and Martinique | Through study completion, an average of 6 years
  Number of new cases per year.

SECONDARY OUTCOMES:
Estimate prevalence of the ALS | Through study completion, an average of 6 years
  Determine the total number of case of ALS diagnosed in Guadeloupe and Martinique on the duration of the study
Clinical criteria of SLA | Through study completion, an average of 9 years
  General, neurological, digestive clinical examination and cardiorespiratory complete and the realization of the score " ALS funtional rating scale "
Study the genetic factors of the ALS | Through study completion, an average of 9 years
  Search for transfers of genes TARDBP, VCP, SOD1:
  According to the genealogical data, we shall target the possible family forms to test at these patient's the various genes known and involved in the disease (transfers of the gene SOD1 (21q22.11), of the gene TARDBP (1p36.22) coding the protein TAR DNA-binding protein 43 (TDP-43) and of the gene VCP (9p13.3) coding for the protein Valosin Containing Protein).
  For the sporadic cases the analysis of these genes will be realized on the whole studied population.
  For the family cases the genetic study will be spread in the whole family.

CONTACTS AND LOCATIONS:
Overall Officials: Annie LANNUZEL, Professor, Neurological, Study Director — Hospital University Center of Pointe-à-Pitre
Locations (2):
- Hospital University Center of Pointe-à-Pitre, Pointe-à-Pitre, Guadeloupe
- Hospital University Center of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No